CLINICAL TRIAL: NCT02006043
Title: A Phase II, Open, Single Arm Trial to Evaluate Erlotinib Efficacy and Safety as the 2nd/3rd Line Treatment in Advanced or Recurrent NSCLC With EGFR Wild Type and Without C-met Expression
Brief Title: Evaluate Erlotinib Efficacy and Safety as the 2nd/3rd Treatment in NSCLC With EGFR M(-) and C-met(-)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Zhang (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28941
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib 150mg/day taken orally (Experimental): Erlotinib 150mg/day taken orally until disease progression or intolerable toxicities
  Interventions: Drug: Erlotinib 150mg

INTERVENTIONS:
Drug: Erlotinib 150mg

SUMMARY:
evaluate Erlotinib efficacy and safety as the 2nd/3rd line treatment in advanced or recurrent NSCLC with EGFR wild type and without c-met expression

DETAILED DESCRIPTION:
In this phase II, open, single arm study, it will be evaluated of the efficacy and safety of erlotinib in 2nd/3rd line of EGFR WT and c-Met negative advanced NSCLC.The treatment goes as follows:Erlotinib 150mg/day taken orally until disease progression or intolerable toxicities.The primary end point of the study was 6 months PFS rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytological documented metastatic (stage IV) or recurrent NSCLC
2. Measurable disease must be characterized according to the response evaluation criteria in solid tumors(RECIST1.1) criteria
3. Must have at least one prior platinum-based chemotherapy regimen for advanced NSCLC and now exhibit progressive disease (PD), and must have recovered from any serious treatment related toxicity
4. Neither with EGFR mutation nor c-met expression on Ventana Benchmark instrument(Met negative expression definition: ≥50% of the cells do not stain or stain with weak intensity (clinical score 0 or 1+) )
5. ECOG Performance Status 0 ~2
6. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
7. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases.
8. Male or female.
9. Age ≥ 18 years and ≤75 years
10. Written (signed) informed consent. Able to comply with study and follow-up procedures.

Exclusion Criteria:

1. Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
2. Received treatment with any other investigational agent, or participated in another clinical trial, with the following exceptions.

   * Chemotherapy-only trials are permitted (if completed≧ 28 days prior to receiving the first dose of study drug).
   * Previous adjuvant or neo-adjuvant treatment for nonmetastatic disease is permitted if completed ≥ 6 months before receiving the first dose of study drug; c)Prior surgery is permitted if performed ≥ 4 weeks before receiving the first dose of study drug and the patient is fully recovered.
   * Prior localized radiotherapy is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented, and provided it has been completed ≥ 4 weeks before receiving the first dose of study drug.
   * Participation in a methodological or observational study in which no investigational agent was given
3. Patients who have brain metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation; previously diagnosed and treated CNS metastases or spinal cord compression without evidence of stable disease (clinically stable imaging) for at least 2 months
4. History of another malignancy in the last 5 years with the exception of the following:

   * Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted.
   * Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
5. Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating oncologist and the ophthalmologist.
6. Any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any study medication or that might affect the interpretation of the results or render the subject at high risk from treatment complications.
7. Female subject who is pregnant or breast-feeding
8. Any unstable systemic disease
9. Hypersensitivity to erlotinib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
6 months PFS rate | at when last patient enrolled 6 months

SECONDARY OUTCOMES:
overall survival, OS | at when last patient enrolled 18 months
objective response rate, ORR | at when last patient enrolled 18 months

OTHER OUTCOMES:
the quality of life of patients | at when last patient enrolled 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-Sen University cnacer center, Guangzhou, Guangdong
  - Guangxi Medical University cancer center, Nanning, Guangxi